CLINICAL TRIAL: NCT03599050
Title: Training in the 21st Century: Using Virtual Role-Plays to Improve Nurse Communication for Medication Adherence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 18-01003
Record Dates: First submitted 2018-07-17; First posted 2018-07-26 (Actual); Last update posted 2022-02-14 (Actual); Status verified 2022-01

CONDITIONS: High Blood Pressure; Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Communication Simulation (Experimental): Nurses will use simulation over 12 weeks while fidelity is monitored using the NIH Behavior Change Consortium Treatment Fidelity Guidelines.
  Interventions: Behavioral: Audiotaped Counseling Session

INTERVENTIONS:
Behavioral: Audiotaped Counseling Session — Patients and nurses will complete audio taped counseling session at least 3 months following the baseline visit. Patients will rate quality of nurse communication skills

SUMMARY:
This study will utilize a three-phase approach that is informed by a theory-driven implementation framework to: 1) conduct a needs analysis in order to identify individual-, health care team-, and practice-level barriers and facilitators to conducting adherence counseling in safety-net primary care practices; 2) develop a virtual communication simulation designed to improve the quality of adherence counseling by allowing nurses repeated opportunities to practice discussing medication adherence with virtual patients; and 3) conduct a pilot study to evaluate the feasibility, acceptability and preliminary efficacy of the simulation on changes in: a) nurses' collaborative communication skills, b) medication adherence, and c) reduction in BP in a sample of 20 patients with uncontrolled hypertension (HTN) who are non-adherent to their medications.

ELIGIBILITY:
Inclusion Criteria:

* PCPs and nurses will be enrolled if they fulfill the following criteria:

  1. male or female healthcare provider (MD/DO, NP, and Registered Nurse) practicing at the clinic
  2. age 18 years or older.

No exclusions will be made based on provider race/ethnic origin. We will oversample males to examine differential communication skills based on gender.

* Patient eligibility criteria include:

  1. receiving care at the participating clinic
  2. having uncontrolled HTN (BP>140/90 mmHg) at two visits in the past year
  3. being prescribed at least one antihypertensive medication and are non-adherent
  4. are ≥age 18 years
  5. fluent in English

Exclusion Criteria:

* Unable to give consent
* Have a diagnosis of cognitive dysfunction or significant psychiatric comorbidity,
* Participating in another HTN-related study.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2020-05-04 (Actual); Study Completion 2020-05-31 (Actual)

PRIMARY OUTCOMES:
Feasibility measured by documenting total available and eligible nurses and patients approached to enroll 1 participant through final study visit | 6 Months
Acceptability measured by % of nurses who complete the simulation | 6 Months

CONTACTS AND LOCATIONS:
Overall Officials: Antoinette Schoenthaler, MD, Study Director — NYU Langone Health
Locations (1):
- NYU School of Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices). Will be used for secondary data analysis approved by the investigator
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 3 months and ending 5 years following article publication.
Access Criteria: Researchers who provide a methodologically sound proposal.